CLINICAL TRIAL: NCT05784714
Title: Development of a Geographical Momentary Assessment Informed Trauma Intervention to Improve ART Adherence and Viral Suppression in Violence-Affected Persons Living with HIV
Brief Title: NOLA GEM: Feasibility and Acceptability of an MHealth Intervention for Violence-affected PLWH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R34AA02896m
Record Dates: First submitted 2023-02-15; First posted 2023-03-27 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-08

CONDITIONS: HIV; Mental Health; Substance Use
Keywords: Adherence; mHealth; Care engagement
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): This arm will include daily diary assessment and GPS phone tracking, access to psychoeducational modules, skills practice, and tools to help with coping and stress reduction. Enhancements include geofencing alerts for risky environments; progress tracking and feedback reports; self-initiated tool engagement (e.g. push button to engage in coping exercise), robust JITAI programming that recommends skills for participants to use in the moment based on daily diary responses, positive mood building exercises, and support.
  Interventions: Behavioral: NOLA GEM
- GEMA (No Intervention): This arm will include daily diary and phone tracking. Participants in this arm will also respond to daily diary assessments twice daily but will not receive the psychoeducation interactive components such as tracking and feedback, alerts, or capacity to send alerts that connect them to tools. This arm will have access to resources.

INTERVENTIONS:
Behavioral: NOLA GEM — This is a mobile application that has 6 psychoeducational sessions and related skills, local resources, and a way for participants to track their progress. Further information is in the arm descriptions.
  Arms: Intervention

SUMMARY:
The objective of the proposed research is to conduct formative work to develop, pilot and refine a smartphone delivered intervention for violence affected people living with HIV utilizing a novel spatial-temporal methodology, geographical ecological momentary assessment (GEMA), to first identify the activity spaces and daily psychosocial experiences (mental health symptoms, substance use, self-efficacy, coping) impacting adherence and viral suppression, and apply them to intervention. Guided by an ecological perspective, the investigators will adapt Living in the Face of Trauma to a mobile platform with GEMA informed intervention targets. The resulting app shall be referred to as NOLA GEM. Our long-term goal is delivering accessible interventions informed by daily experiences that affect health for PLWH. The investigators will test feasibility, acceptability and preliminary efficacy of the GEMA-informed NOLA GEM app against GEMA alone on adherence and care, and secondary outcomes of mental health and substance use.

ELIGIBILITY:
Inclusion Criteria:

* Having a reported HIV infection and being on ART.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Adherence | 30 day post-assessment
  Self report taking all HIV-related medication and treatment in past 30 days
Viral Load | 90 days post assessment
  Self report last blood draw was under 50 copies of HIV/mL in past 90 days
Care Engagement | 90 days post assessment
  Self report % of missed appointments in past 90 days
Care Engagement | 30 days post assessment
  HIV Treatment Adherence Self-Efficacy Scale; 0-120; higher score means more self-efficacy for care engagement
Acceptability of intervention | 30 day post-assessment
  User Experience Questionnaire-Short Form
Acceptability of intervention | 30 day post-assessment
  Net Promotor Score; 0-10; higher score means more likely to recommend to a friend
Feasibility of intervention | 30 day post-assessment
  App usage paradata
Feasibility of intervention | 30 day post-assessment
  Participation rates

SECONDARY OUTCOMES:
PTSD | 30 day post-assessment
  PTSD Checklist for DSM-5; higher scores indicate higher levels of PTSD symptomology
Depression, anxiety | 30 day post-assessment
  Hospital Anxiety Depression Scale; 0-21; higher scores indicate higher levels of anxiety and/or depression
Stress | 30 day post-assessment
  Study generated daily stressors severity checklist
Stress | 30 day post-assessment
  Perceived Stress Scale 4; 0-16; higher score is correlated to more stress
Coping | 30 day post-assessment
  Brief-COPE; higher scores indicate higher levels of emotion focused, problem focused, and avoidant coping styles
Coping | 30 day post-assessment
  adapted Coping Self-Efficacy Scale; higher score means more coping self-efficacy
Substance use | 30 day post-assessment
  Adapted Addiction Severity Index
Substance use | 30 day post-assessment
  Alcohol Use Disorders Identification Test-C; 0-12; higher score indicates more problematic drinking

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Access Health Louisiana, New Orleans, Louisiana
  - Women With A Vision, New Orleans, Louisiana
  - CrescentCare, New Orleans, Louisiana
  - Institute of Women & Ethnic Studies, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gasik RE, Skeen SJ, Tokarz S, Theall KP, Clum GA. Outcomes of a Pilot Mobile App Just-in-Time-Adaptive-Intervention Supporting Coping Skills in Trauma Affected People with HIV. AIDS Behav. 2026 Jan 23. doi: 10.1007/s10461-026-05032-6. Online ahead of print. PMID 41575709
- [Derived] Skeen SJ, Tokarz S, Gasik RE, Solano CM, Smith EA, Sagoe MB, Hudson LV, Steele K, Theall KP, Clum GA. A Trauma-Informed, Geospatially Aware, Just-in-Time Adaptive mHealth Intervention to Support Effective Coping Skills Among People Living With HIV in New Orleans: Development and Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 24;12:e47151. doi: 10.2196/47151. PMID 37874637